CLINICAL TRIAL: NCT06786104
Title: A Multisite RWCT Comparing the Effectiveness of a Goals of Care Video and Navigator Intervention, the VIDEO-PEDS Experience, Versus Usual Care in Pediatric Cancer
Brief Title: Video Inspired Discussions About Ethical Outcomes in Pediatrics
Acronym: VIDEO-PEDS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Dartmouth-Hitchcock Medical Center (Other); Dana-Farber Cancer Institute (Other); Yale University (Other); Emory University (Other); Children's Healthcare of Atlanta (Other); University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Joanne Wolfe, MD, MPH, Chief of Pediatrics, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 24-313; 1UG3CA286852-01A1 (NIH)
Record Dates: First submitted 2025-01-07; First posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Pediatric Cancer
Keywords: Advanced Care Planning; Palliative Care; End of Life
MeSH Terms: conditions — Neoplasms; Death | interventions — Focus Groups

STUDY DESIGN:
Intervention Model Description: The initial development and pilot phase is not randomized and the latter RWCT phase is 1:1 parallel randomized arms.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- UH3 RWCT Arm - Intervention (Experimental): This group will receive the VIDEO-PEDS intervention.
  Interventions: Other: VIDEO-PEDS
- UH3 RWCT Arm - Control (No Intervention): This group will receive usual care until the 9-month wait period expires.
- UG3 Pilot Intervention (Other): This group will receive the 3-month pilot version of the VIDEO-PEDS intervention.
  Interventions: Other: VIDEO-PEDS pilot
- UG3 Focus Group (Other): This group will participate in the virtual parent focus groups.
  Interventions: Other: Focus Group

INTERVENTIONS:
Other: VIDEO-PEDS — Following enrollment, parents will receive a link to view the refined video decision aid that is designed to prompt parents to think about their goals of care for their child with cancer, and then to react by engaging in communication with a trained member of the research team called the Navigator and eventually their clinical team over the course of the 9-month study duration.
  Arms: UH3 RWCT Arm - Intervention
Other: VIDEO-PEDS pilot — This is the 3-month pilot version of the intervention, which will be further developed for the eventual RWCT.
  Arms: UG3 Pilot Intervention
Other: Focus Group — Parents will view the Video aid and provide fascilitated feedback in an audio-recorded virtual group setting.
  Arms: UG3 Focus Group

SUMMARY:
The goal of this clinical trial is to learn if the VIDEO-PEDS intervention works to improve Goals of Care communication between clinicians and parents of children with cancer.

The main questions it aims to answer are:

Does the intervention improve Goals of Care documentation? Does it improve patient outcomes (including less invasive preferences for resuscitation and interventions, less hospital utilization, and more palliative care and hospice use)? Does it improve parent outcomes (including health satisfaction and feeling heard and understood per survey scores)?

DETAILED DESCRIPTION:
Background

Parents of children with advanced cancer often face challenging decisions about goals of care (GOC) amidst high stress and limited understanding of medical interventions. Despite evidence that early and informed GOC discussions improve end-of-life experiences and align care with family values, such conversations remain infrequent in pediatric oncology. Barriers such as communication gaps, literacy challenges, and cultural differences exacerbate disparities, particularly among African American, Hispanic, and rural populations. The Video Images about Decisions for Ethical Outcomes in Pediatrics (VIDEO-PEDS) trial aims to address these gaps through an innovative video-based intervention. Similar interventions were effective in an adult cancer population.

Aims

1. To refine and finalize a theory-based video decision aid tailored to parents of children with advanced cancer.
2. To evaluate the feasibility, acceptability, and preliminary impact of the intervention through a pilot study.
3. To conduct a randomized waitlist-controlled trial (RWCT) assessing the effectiveness of the intervention in improving GOC communication and documentation.

Design

This study will be conducted in two phases:

1. Pilot Study

   * Design: A mixed-methods study to test the feasibility and acceptability of the intervention among 27 parents (9 per site). Focus groups with 36 parents (12 per site) will be conducted in English and Spanish. Clinician providers will be interviewed.
   * Purpose: To refine the intervention and ensure its appropriateness for the larger trial.
2. Randomized Waitlist-Controlled Trial (RWCT)

   * Design: A multicenter, parallel-group RCT with a waitlist control.
   * Purpose: To evaluate the impact of the intervention on GOC documentation and patient- and parent-centered outcomes.

Setting

The study will take place across three diverse healthcare systems:

1. Dana-Farber Cancer Institute/Boston Children's Hospital
2. Children's Healthcare of Atlanta/Aflac Cancer Center
3. University of Alabama at Birmingham These sites were selected because of their robust pediatric oncology programs and diverse patient populations, including African American, Hispanic, and rural families.

Participants/Subjects

1. Pilot Study:

   Parents of 27 children (9 per site) aged 0-12 years with cancer will be recruited to test the intervention.
2. RWCT:

   * A total of 504 parents (168 per recruitment cycle across three cycles) will be enrolled.
   * Stratification will ensure representation of African American, Hispanic, and rural populations.

Interventions

1. Pilot Study:

   * Intervention: A video decision aid coupled with structured conversations facilitated by trained Navigators. The video provides education about GOC, focusing on values-based decision-making and specific interventions (e.g., CPR, intubation).
   * Duration: Parents will view the video and engage in one or more conversations with the Navigator over three months.
2. RWCT:

   * Intervention: Refined video decision aid with Navigator-led discussions over a nine-month period.
   * Control: Usual care, with the intervention provided to the waitlist control group after nine months.

Methods Patients will be screened from oncology patient lists at the three enrolling sites. A research assistant will complete an eligibility checklist for all meeting general criteria after an initial screening. For those potentially eligible, an eligibility checklist will be reviewed by a site PI and validated (eventually through REDCap). Once deemed eligible, an opt-out email is sent to the primary clinician for permission to approach. Invitations will then be sent by mail or email, followed by an in-person or phone approach. Prospective verbal informed consent will be obtained from the parents who choose to participate. Participation then involves viewing the Video. Video cards (inexpensive disposable devices) may be provided to reduce barriers to participation. Following the viewing, an extensively trained Navigator from the research team will discuss the goals of care broadly with the parent throughout the study duration, prompting engagement with the primary oncologist.

Development Phase:

* Parent focus groups led by site PIs will be held in English and Spanish via Zoom and audio recorded. The video will be shown and discussed following a semi-structured guide.
* The video will be refilmed to incorporate feedback from the focus groups.
* Workflows will be refined and study infrastructure will be developed further for the next phase.

Pilot Study:

o An abbreviated 3-month version of the intervention will be tested, including pre- and post-study surveys.

RWCT:

The investigators will conduct a large, pragmatic, randomized, waitlist-controlled trial (RWCT). The investigators will conduct three cycles of nine months. Thus, over the course of 27 months, three cycles of unique patients will be randomized (9 months per cycle x 3 cycles = 27 months). The recruitment period is 36 months to account for the last nine months of intervention for Waitlist-Controls in the last cycle. At the start of each of the three cycles, the investigators will ask each health system to curate and finalize a list of all eligible patients. For each cycle, one-third of the total 504 (i.e., N=168) will be randomized in 1:1 assignment, stratified by health system and demographic characteristics (African American, Hispanic, and rural) to Waitlist-Control or GOC Video Intervention.

A subgroup of 136 parents (total) will be asked to complete a survey via REDCap. These parents will be evenly divided between the two arms of the study and the three study sites. Participants will receive a self-administered survey via email/mailing at the beginning of a nine-month period and again at the end.

A subgroup of 12 parents (total) will be asked to complete an audio-recorded exit interview. The investigators will ask parents to comment on the perceived usefulness of the intervention, whether anything was learned, and how communication may have changed with the participant's clinicians since the intervention.

A subgroup of 25 parents (total) will have the Navigator conversation audio-recorded for intervention fidelity. A subset of these will be transcribed and further analyzed.

Stakeholder Interviews will be conducted with 18 clinicians (6 per site) including key clinical leaders of services.

Data Analysis:

* Mixed-methods process evaluation will use the RE-AIM framework to assess implementation.
* Descriptive statistics will be used for feasibility outcomes (e.g., recruitment, and retention rates).
* Comparative analysis of primary and secondary outcomes between intervention and control groups using intention-to-treat principles.
* Natural Language Processing technology will be used to identify outcomes in the EHR.

Outcomes

While more detail on Outcomes exists in that section, the primary outcome for the RWCT is the presence of GOC documentation in the EHR. Secondary outcomes include:

* Implementation outcomes: Feasibility, acceptability, and fidelity of the intervention.
* Parent-reported outcomes: Satisfaction with communication, perceived knowledge, and decisional certainty.
* Patient outcomes: Location of care at the end of life, alignment of care with stated goals.

Exploratory analyses will examine subgroup effects among African American, Hispanic, and rural participants, as well as the cost-effectiveness and scalability of the intervention.

ELIGIBILITY:
Inclusion Criteria:

Patient

* Age 0-12 years
* Diagnosed with any type or stage of cancer
* Receiving cancer directed treatment

Parent

* Decision maker for the child.
* Biological parent, step-parent, legal guardian (e.g., adoptive parent), or grandparent with medical consent authority.
* Has a child meeting the child inclusion criteria listed above.
* Able to communicate in English or Spanish (the languages of the video decision aids).

Exclusion Criteria:

Patient

* Not receiving primary medical care from the cancer clinic (e.g., second-opinion consultations only)
* Already referred to and fully consulted by the palliative care team
* Prognosis of less than a 2-month life expectancy

Parent

* Visually impaired beyond 20/200 corrected and unable to view the video (note: hearing impaired is not an exclusion as the videos are closed captioned).
* Psychological state not appropriate for GOC discussions, as determined by the primary oncologist per the opt-out.
* Participants who do not speak English or Spanish

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 567 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2030-01-15 (Estimated); Study Completion 2030-04-15 (Estimated)

PRIMARY OUTCOMES:
Goals-of-Care Discussion | At the end of Cycles 1, 2, and 3 (each cycle is 9 months)
  Percentage of parents who held conversations with their medical team about goals, values, or priorities for treatment and outcomes as per documentation in the medical record.
Code Status Limitation | At the end of Cycles 1, 2, and 3 (each cycle is 9 months)
  Percentage of parents who communicate limitations to cardiopulmonary resuscitation and intubation with their medical team as per documentation in the medical record.
Palliative Care | At the end of Cycles 1, 2, and 3 (each cycle is 9 months)
  Percentage of parents who mention a visit with a specialty palliative care clinician, mention of specialist palliative care discussion, or patient preferences regarding seeing a palliative care clinician to their medical team as per documentation in the medical record.
Time-Limited Trial | At the end of Cycles 1, 2, and 3 (each cycle is 9 months)
  Percentage of parents who engage in conversations with their medical team about the use of a treatment or procedure for a set amount of time with a pre-defined goal and plan related to the outcome at the end of the trial as per documentation in the medical record.

SECONDARY OUTCOMES:
Acceptability themes from qualitative data | 2 years
  For the development phase, qualitative group interviews will yield information about participant preferences. For the pilot phase, qualitative individual interviews will yield information about participant preferences after a 3-month study duration.
Feasibility by % of parents | 2 years
  Feasibility will be assessed as ability to identify, recruit, and retain participants as a percentage. 70% of those screened should be eligible for approach after the Validation and Opt-out Steps. 70% approached should agree to participate. 70% should complete the study. (<30% should be lost to follow-up or withdraw from the study.)
Parent Satisfaction scores | 2 years
  A parent survey will measure how parents felt heard and understood by the medical team and how satisfied they were with the care received using five validated items from the measure Feeling Heard and Understood and two items from the Survey about Caring for Children with Cancer (SCCC) all answered on a 5-point Likert Scale. Scores range from 0 to 100 with 0 being the lowest satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Angelo Volandes, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (4):
- United States (4):
  - Children's of Alabama at Birmingham, Birmingham, Alabama
  - Children's Hospital of Atlanta, Atlanta, Georgia
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Volandes AE, Zupanc SN, Lakin JR, Cabral HJ, Burns EA, Carney MT, Lopez S, Itty J, Emmert K, Martin NJ, Cole T, Dobie A, Cucinotta T, Joel M, Caruso LB, Henault L, Dugas JN, Astone K, Winter M, Wang N, Davis AD, Garde C, Rodriguez PM, El-Jawahri A, Moseley ET, Das S, Sciacca K, Ramirez AM, Gromova V, Lambert S, Sanghani S, Lindvall C, Paasche-Orlow MK. Video Intervention and Goals-of-Care Documentation in Hospitalized Older Adults: The VIDEO-PCE Randomized Clinical Trial. JAMA Netw Open. 2023 Sep 5;6(9):e2332556. doi: 10.1001/jamanetworkopen.2023.32556. PMID 37695586
- [Background] Snaman JM, Feifer D, Helton G, Chang Y, El-Jawahri A, Volandes AE, Wolfe J. A Pilot Randomized Trial of an Advance Care Planning Video Decision Support Tool for Adolescents and Young Adults With Advanced Cancer. J Natl Compr Canc Netw. 2023 Jul;21(7):715-723.e17. doi: 10.6004/jnccn.2023.7021. PMID 37433434
- [Background] Feifer D, Helton G, Wolfe J, Volandes A, Snaman JM. Adolescents and young adults with cancer conversations following participation in an advance care planning video pilot. Support Care Cancer. 2024 Feb 17;32(3):164. doi: 10.1007/s00520-024-08372-y. PMID 38367086
- [Background] Lindsay ME, de Oliveira S, Sciacca K, Lindvall C, Ananth PJ. Harnessing Natural Language Processing to Assess Quality of End-of-Life Care for Children With Cancer. JCO Clin Cancer Inform. 2024 Sep;8:e2400134. doi: 10.1200/CCI.24.00134. PMID 39265122
- [Background] Johnston EE, Alvarez E, Saynina O, Sanders L, Bhatia S, Chamberlain LJ. Disparities in the Intensity of End-of-Life Care for Children With Cancer. Pediatrics. 2017 Oct;140(4):e20170671. doi: 10.1542/peds.2017-0671. PMID 28963112
- [Background] Lindvall C, Deng CY, Moseley E, Agaronnik N, El-Jawahri A, Paasche-Orlow MK, Lakin JR, Volandes A, Tulsky TAIJA. Natural Language Processing to Identify Advance Care Planning Documentation in a Multisite Pragmatic Clinical Trial. J Pain Symptom Manage. 2022 Jan;63(1):e29-e36. doi: 10.1016/j.jpainsymman.2021.06.025. Epub 2021 Jul 14. PMID 34271146

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-05-01): https://cdn.clinicaltrials.gov/large-docs/04/NCT06786104/Prot_SAP_000.pdf